CLINICAL TRIAL: NCT03438188
Title: Neural Basis of Eating Behavior in Abstinent Smokers
Acronym: SIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, James Loughead, Associate Professor, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 828958
Record Dates: First submitted 2018-02-09; First posted 2018-02-19 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Nicotine Use Disorder
Keywords: Nicotine Addiction; Quitting Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: This is a within-subject cross-over neuroimaging investigation of 3 potential neural mechanisms of increased caloric intake during initial smoking cessation. Eighty smokers will be scanned on 2 occasions: (1) after 4 days of monitored abstinence (biochemically verified), and (2) after 4 days of smoking as usual (order counterbalanced). In addition, 30 healthy non-smokers (matched for sex, age, and education) will complete one period of the study to serve as a baseline comparison group.
Masking Description: Smoking participants will be studding under both smoking as usual and abstinent conditions (crossover) and non-smokers only under "abstinence."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoker Group (Experimental): The smokers group will be scanned on 2 occasions: (1) after a 4 day monitored practice quit attempt (biochemically verified), and (2) after 4 days of smoking as usual (order counterbalanced).
  Interventions: Other: Practice Quit Attempt
- Non-Smoking Comparison Group (No Intervention): Healthy non-smokers will complete one period (comparable to abstinence arm) of the study to serve as a baseline comparison group.

INTERVENTIONS:
Other: Practice Quit Attempt — Smokers will be studied under 2 conditions: smoking as usual and during a 4 day practice quit attempt.
  Arms: Smoker Group

SUMMARY:
The purpose of this research study is to better understand why people gain weight when they quit smoking by examining food intake and changes in brain activity in smokers when they are smoking as usual compared to when they have been deprived of cigarettes (i.e., have not smoked for 4 days) as compared to a non-smoker control group.

DETAILED DESCRIPTION:
Tobacco use and obesity are the two leading causes of preventable deaths. Because these two behaviors share common brain reward mechanisms, reducing one behavior often leads to increases in the other behavior. Behavioral Economic and Incentive Salience models shed much light on this clinical problem. Smoking cessation produces reward dysregulation that can alter the motivational salience of other reinforcers, particularly food. After stopping smoking, smokers increase between-meal snacking, especially foods high in fat and sugar. Increases in caloric intake occur within days of quitting smoking, and are clinically significant. The investigators have also shown that smoking cessation produces working memory deficits and reduces activity in the brain's cognitive control circuits, making it even more difficult to exert self-control over temptations to eat highly rewarding foods. Thus, smokers have a double challenge: food becomes more salient and reinforcing at a time when their neurocognitive resources are compromised.

Neuroimaging can identify mechanisms underlying behavior change beyond self-report and behavioral measures. The proposed functional magnetic resonance imaging (fMRI) study breaks new ground by integrating concepts and tools from the fields of behavioral economics and cognitive neuroscience to accelerate the study of mechanisms underlying PCWG. The investigators will use a previously validated within-subject crossover neuroimaging study design to examine changes in working memory, food salience (cue-induced craving), and food reinforcement processes in the brain after 4 days of smoking cessation (vs. smoking as usual). A non-smoker control group will provide insight into baseline differences from smokers (abstinent and satiated). Caloric intake, the primary outcome, will be assessed using 24-hr. food recalls during each study period. The investigators will assess three parallel pathways including: working memory, food cue reactivity, and food reinforcement at the neural and behavioral levels.

This study will provide new insights about how the brain can constrain or promote the ability of smokers to prevent post cessation weight gain (PCWG) and lead to new interventions that integrate neural and behavioral framework. Support for our predictions would inform testing of novel approaches to prevent PCWG, such as computerized neurocognitive exercise training to increase DLPFC activity and shift activity away from reward sensitive brain networks.

ELIGIBILITY:
Inclusion Criteria

Male and female participants who are between 18 and 45 years of age.

Smoking group - 80 treatment-seeking smokers who self-report smoking at least 10 cigarettes (menthol and/or non-menthol) per day for at least the last 6 months. Smoking status will be confirmed by CO greater than or equal to 8 parts per million (ppm) at the Intake Visit.

Non-smoking group - 30 individuals reporting fewer than 100 lifetime cigarettes and not even a puff of a cigarette for a minimum of 2 years. Smoking status of non-smokers will be confirmed by CO less than 5ppm. They will be matched to the smoker group on age, sex, and education.

Plan to live in the area for the duration of the study (i.e. ~8 weeks/2 months).

Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.

Smokers who wish to make a permanent quit attempt in the next 1-2 months (treatment-seeking), because our prior work suggests that motivated subjects are more sensitive to medication effects on smoking behavior. Using a scale from 0 to 100 (100, being extremely interested), subjects must rate their interest in quitting smoking within the next 1-2 months greater than 50.

Able to communicate fluently in English (i.e. speaking, writing, and reading).

Exclusion Criteria

Subjects who present and/or self-report with the following criteria will not be eligible to participate in the study:

Smoking Behavior

1. Regular use of nicotine-containing products other than cigarettes (e.g. chewing tobacco, snuff, snus, cigars, e-cigs, etc.). Participants agreeing to abstain from using nicotine- containing products other than cigarettes will be considered eligible.
2. Current enrollment or plans to enroll in another research and/or smoking cessation program over the duration of the study (i.e. ~8 weeks/2 months).
3. Anticipated use (within the next ~8 weeks/2 months) of any nicotine substitutes and/or smoking cessation treatments/medications unless provided through the study.
4. Provide a CO breath test reading less than 8 ppm at Intake Visit (smokers) or greater than 5ppm at intake visit (non-smokers).

Alcohol and Drug

1. History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse. Counseling and support groups (e.g. Alcoholics Anonymous and Narcotics Anonymous) will not be considered medical treatment for the purposes of this protocol.
2. Current alcohol consumption that exceeds 25 standard drinks/week.
3. Breath alcohol reading (BrAC) greater than .000 at the Intake Visit.
4. A positive urine drug screen (UDS) for cocaine, opiates, amphetamines, methamphetamines, phencyclidine (PCP), ecstasy (MDMA), barbiturates, benzodiazepines, methadone, and/or oxycodone at the Intake Visit.

Medical

1. Women who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period. Women must agree to use an adequate form of contraception or abstain from sexual intercourse for the duration of the study.
2. Current treatment of cancer or diagnosed with cancer (except basal or squamous-cell carcinoma not treated with chemotherapy and/or radiation) in the past 6 months.
3. Poorly controlled, brittle, or pump-dependent Type I diabetes.
4. Current peptic ulcer bleeding.
5. Active hepatitis or poorly controlled kidney and/or liver disease.
6. Serious or unstable disease within the past 6 months. Notable diseases will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
7. Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing proper completion of the study procedures. Notable impairments will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
8. Applicable food allergies or disorders:

   * Galactosemia a
   * Notable milk allergy (lactose intolerant participants may proceed unless they experience severe symptoms) b
   * Notable soy allergy c
   * Peanut allergy d a,b,c Boost® Original Very Vanilla Nutritional Shake: Contains milk and soy ingredients. Suitable for Lactose Intolerance.

     1. b,c,d M&M's® (Milk Chocolate): Contains milk and soy ingredients (MAY CONTAIN PEANUTS) Lay's® Classic Potato Chips (Gluten Free): Potatoes, vegetable oil, and salt

Psychiatric

1. Current diagnosis of major depression. Subjects with a history of major depression, in remission for 6 months or longer (may be stable on antidepressant medications), are eligible.
2. Lifetime history of a suicide attempt.
3. Lifetime history of schizophrenia, psychosis, and/or bipolar disorder.
4. Current diagnosis of Attention Deficit/Hyperactivity Disorder (ADHD).
5. Current diagnosis of bulimia, anorexia nervosa or binge eating.

Medication

Current use or recent discontinuation (within the last 14 days) of:

1. Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin SR, Chantix).
2. Benzodiazepines and/or Barbiturates.
3. Anti-psychotic medications.
4. Prescription stimulants (e.g., Provigil, Ritalin, Adderall).
5. Systemic steroids.
6. Medications for the use of addiction treatment.

   Current use of:
7. Nicotine replacement therapy (NRT).
8. Heart medications such as digoxin, quinidine, and nitroglycerin.

   Daily use of:
9. Opiate-containing medications for chronic pain.
10. Inhaled corticosteroids.

Subjects will be instructed to refrain from using any study-prohibited drugs/medications (both recreational and prescription) throughout their participation in the study. After final eligibility is confirmed, subjects who report taking contraindicated medication(s) over the course of the study period may only remain eligible if the Study Physician and Principal Investigator determine that the contraindicated medication(s) do/did not significantly impact the study design, data quality, and/or subject safety and welfare. Subjects are permitted to take necessary prescription medications not included within the exclusion list during the study.

General Exclusion

1. Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator and/or Study Physician.
2. Participation in a dietary program within the past 30 days.
3. Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator and/or Study Physician. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.
4. Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/or Study Physician. Subjects may be deemed ineligible at any point throughout the study.
5. Low or borderline intellectual functioning - determined by receiving a score of less than 85 on the Shipley Institute of Living Scale (SILS), which correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated IQ Test.

fMRI Exclusion Criteria

1. History of claustrophobia.
2. Being left-handed.
3. Lifetime history of stroke.
4. Having a cochlear implant or wearing bilateral hearing aids.
5. History of notable head trauma. Although notable head trauma is typically defined as being knocked unconscious for a period of three minutes or longer, notable head trauma will be evaluated on a case-by-case basis by the appropriate personnel prior to an eligibility decision, considering exceptions can be made based on the nature and severity of the trauma.
6. History of brain or spinal tumor.
7. Pacemakers, certain metallic implants or objects, or presence of metal in the eye as contraindicated for MRI.
8. Any circumstances (e.g., exclusionary metal implants, certain dental work, and/or physical impairments) and/or conditions that may interfere with MRI and MRI-related study visit procedures. All potential exclusionary circumstances and/or conditions will be evaluated on a case-by-case basis by the appropriate personnel prior to an eligibility decision.
9. History of gunshot wounds. Injuries from BB guns will be evaluated on a case-by-case basis by the appropriate personnel prior to an eligibility decision.
10. History of epilepsy and/or recurrent or uncontrolled seizures.
11. Weight greater than 250 lbs at Intake Visit or self-reported at phone screen. If a participant weighs less than or equal to 250 lbs at Intake, but presents with a weight greater than 250 lbs at either Scan 1 and/or Scan 2, the participant may be permitted to proceed with the scan as long as the participant's weight does not exceed 300 lbs.
12. A positive urine drug screen (UDS) for cocaine, opiates, amphetamines, methamphetamines, phencyclidine (PCP), ecstasy (MDMA), barbiturates, benzodiazepines, methadone, and/or oxycodone at intake or either Scan Visit.
13. A BrAC greater than 0.000 at intake or either Scan Visit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Loughead, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Smoking Then Abstinent Group: The Smoking then Abstinent Group group will be scanned on 2 occasions:(1) after 4 days of smoking as usual, and (2) after a 4-day monitored practice quit attempt (biochemically verified).
- Abstinent Then Smoking Group: The Abstinent then Smoking Group group will be scanned on 2 occasions: (1) after a 4-day monitored practice quit attempt (biochemically verified), and (2) after 4 days of smoking as usual.
Period: Scan 1(Smoking, Abstinent or Non-smoker)
Arm/Group | Smoking Then Abstinent Group | Abstinent Then Smoking Group | Non-Smoking Comparison Group
Started | 25 | 26 | 31
Completed | 17 | 18 | 27
Not Completed | 8 | 8 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Lost to Follow-up | 4 | 3 | 2
Not completed — change in eligibility | 3 | 4 | 1
Period: Washout Period (Smoking or Abstinent)
Arm/Group | Smoking Then Abstinent Group | Abstinent Then Smoking Group | Non-Smoking Comparison Group
Started | 17 | 18 | 0 (Non-smoking Group received one scan.)
Completed | 14 | 14 | 0 (Non-smoking Group received one scan.)
Not Completed | 3 | 4 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — change in eligibility | 3 | 2 | 0
Period: Scan 2 (Smoking or Abstinent)
Arm/Group | Smoking Then Abstinent Group | Abstinent Then Smoking Group | Non-Smoking Comparison Group
Started | 14 | 14 | 0 (Non-smoking Group received one scan.)
Completed | 14 | 14 | 0 (Non-smoking Group received one scan.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoking Then Abstinent Group | Abstinent Then Smoking Group | Non-Smoking Comparison Group | Total
Number analyzed (Participants) | 25 | 26 | 31 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.38 (14.31) | 46.40 (13.68) | 39.65 (14.86) | 43.74 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 20 | 42
  Male | 15 | 14 | 11 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 2 | 10
  Not Hispanic or Latino | 22 | 21 | 29 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 16 | 18 | 49
  White | 5 | 5 | 8 | 18
  More than one race | 4 | 2 | 5 | 11
  Unknown or Not Reported | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Abstinence Induced Change in Task BOLD Signal Change
Description: The primary outcome measure is change in BOLD signal for the Food Cue-Induced Craving primary regions of interest for the BOLD fMRI analysis are anterior cingulate gyrus (ACC), Insula, Ventral Striatum (VS), and orbital frontal cortex (OFC). For the Working Memory N-Back Task the primary regions of interest for the BOLD analysis will be dorsal lateral prefrontal cortex (DLPFC) and posterior cingulate gyrus (PCC).
Time Frame: BOLD fMRI is collected on days 4 and 32 of protocol
Population: The smoking and abstinent fMRI session population is comprised of all smokers completing two fMRI sessions. The healthy comparison group is composed of all control group participants completing one fMRI scan.
Measure: Mean (Standard Deviation); unit: percentage of signal change
Groups:
- Smoking fMRI Session: The Smoking scan on takes place after 4 days of smoking as usual.
- Abstinent fMRI Session: The Abstinent scan takes place after a 4-day monitored practice quit attempt (biochemically verified).
Arm/Group | Smoking fMRI Session | Abstinent fMRI Session | Non-Smoking Comparison Group
Number analyzed (Participants) | 28 | 28 | 27
percentage of signal change
  Food Induced Craving (ACC) | 0.000 (0.250) | -0.014 (0.233) | 0.027 (0.215)
  Food Induced Craving (Left Insula) | 0.051 (0.252) | -0.011 (0.254) | 0.055 (0.247)
  Food Induced Craving (Right Insula) | 0.057 (0.263) | -0.013 (0.266) | 0.057 (0.246)
  Food Induced Craving (Left VS) | -0.057 (0.359) | 0.062 (.559) | 0.010 (0.497)
  Food Induced Craving (Right VS) | -0.050 (0.330) | 0.053 (0.625) | 0.014 (0.368)
  Food Induced Craving (OFC) | 0.015 (0.227) | 0.034 (0.338) | 0.104 (0.341)
  N-Back Task (left dorsal lateral prefrontal cortex) | 0.211 (0.202) | 0.180 (0.237) | 0.211 (0.378)
  N-Back Task (right dorsal lateral prefrontal cortex) | 0.231 (0.214) | 0.196 (0.239) | 0.243 (0.406)
  N-Back Task (posterior cingulate cortex) | -0.081 (0.202) | -0.096 (0.215) | -0.142 (0.273)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 3 three-month period (2 months in person with 1-month phone follow-up).
Description: Adverse event reporting includes the total number of participants by intervention, whereas the Participant Flow module reports participants by order of administration of intervention. For total at-risk in adverse event tables, the participants for the two counterbalanced orders are summed (e.g. 25 (smoking then abstinent)+26 (abstinent then smoking) = 51 total) for a total at-risk by intervention.
Groups:
- Smoking as Usual (4 Days): The Smoking session takes place after 4 days of smoking as usual.
- Washout (2 Weeks): Washout occurs between scan 1 and scan 2 for the smoking group only.
- Abstinent (4 Day Practice Quit Attempt): The Abstinent session takes place after a 4-day monitored practice quit attempt (biochemically verified).
- Non-Smoking Comparison Session: Healthy non-smokers will complete one period (comparable to abstinence arm) of the study to serve as a baseline comparison group.
Arm/Group | Smoking as Usual (4 Days) | Washout (2 Weeks) | Abstinent (4 Day Practice Quit Attempt) | Non-Smoking Comparison Session
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/31 | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/31 | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 3/51 | 0/31 | 2/28 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoking as Usual (4 Days) (N=51) | Washout (2 Weeks) (N=31) | Abstinent (4 Day Practice Quit Attempt) (N=28) | Non-Smoking Comparison Session (N=31)
incidental finding (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — MRI Technologist reported possible incidental finding during MRI. Scans were evaluated by Study Physician who found nothing significant and no follow-up was required.
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — A participant reported feeling fatigued and weak.
Back Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — A participant experienced back pain during MRI scan.
tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — A participant had oral surgery for an impacted tooth.
Swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Participants had minor injuries with swelling. Accidents were unrelated to study procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03438188/Prot_SAP_000.pdf